CLINICAL TRIAL: NCT01964638
Title: Comparative Analysis of Software-based MRI-Ultrasound Image Fusion Against Cognitive Targeting of Multi-Parametric MRI Findings With Prostate Biopsy
Brief Title: Use of Multi-Parametric MRI With Prostate Biopsy for Cancer Diagnosis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Principal Investigator, Samir Taneja, MD, Co-Director, Smilow Comprehensive Prostate Cancer Center, NYU Langone Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S12-01613
Record Dates: First submitted 2013-10-10; First posted 2013-10-17 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-10

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Prostate Biopsy; Targeted Biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Targeted Biopsy (Other): Men being evaluated for prostate cancer based upon standard of care clinical parameters (e.g. elevated PSA levels, abnormal DRE, mpMRI) will be considered for enrollment. Men who have undergone prostate mpMRI that has revealed an area(s) of suspicion for prostate cancer are eligible for enrollment. All men enrolled in the study undergo fusion targeted biopsy, visual estimation biopsy, and systematic biopsy. As a result the study includes a single arm with direct comparison of biopsy techniques.
  Interventions: Procedure: Targeted Biopsy

INTERVENTIONS:
Procedure: Targeted Biopsy

SUMMARY:
This is a prospective single center trial to examine the rates of cancer diagnosis when using computerized software to target suspicious lesions within the prostate identified on mpMRI. The primary evaluation involves comparing the rate of cancer diagnosis when using software-based MRI-Ultrasound image fusion guided biopsy to sample mpMRI findings to the use of visual guided biopsy (cognitive or mental targeting) of the same target. The hypothesis being tested is that fusion guided biopsy will increase detection prostate cancer within mpMRI findings as compared to visual guided biopsy of these areas

ELIGIBILITY:
Inclusion Criteria:

* No previous diagnosis of adenocarcinoma of the prostate
* No contraindication to prostate biopsy (e.g. coagulopathy, medical condition prohibiting abstinence from anti-platelet or anticoagulation therapies, anatomical considerations, anatomical considerations)
* Active urinary tract infection

Exclusion Criteria:

* Prior pelvic radiotherapy
* Prior androgen deprivation therapy
* Evidence urinary tract infection or significant urinary retention
* Prostate instrumentation (e.g. prostate biopsy, transurethral prostate procedure) within 2 months prior to mpMRI.
* Contraindication to MRI (severe claustrophobia, indwelling metallic objects incompatible with MRI, pacemaker)

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2012-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of rates of prostate cancer diagnosis | One week after biopsy
  The primary endpoint of the study is the evaluation of the rates of prostate cancer diagnosis using software based MRI-TRUS imaging fusion targeting of mpMRI lesions as compared to cognitive co-registration and targeting of mpMRI lesions.

SECONDARY OUTCOMES:
Evaluation of Rate of cancer diagnosis using targeted biopsy | One week after biopsy
  The secondary endpoint of the study is the evaluation of the rate of cancer diagnosis using targeted biopsy (software or cognitive targeting) as compared to standard of care prostate biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Samr S Taneja, MD, Principal Investigator — Co-Director, Smilow Comprehensive Prostate Cancer Center
Locations (1):
- NYU Smilow Prostate Cancer Center, New York, New York, United States